CLINICAL TRIAL: NCT06862362
Title: China Chronic Cough Cohort Study
Brief Title: China Chronic Cough Registry: a Multicenter, Prospective, Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kefang Lai, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: ES-2025-K005-01
Record Dates: First submitted 2025-02-23; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Cough (CC)
Keywords: chronic cough; registry; clinical data; biosample
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — sputum cells, sputum supernatant, PBMC, serum, urine specimens, airway mucosa and bronchoalveolar lavage fluid (BALF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with chronic cough

SUMMARY:
The aim is to establish a national clinical database and biobanks for chronic coughers. Through real-world chronic cough case registry and follow-up studies, we will explore the clinical phenotypes and molecular subtypes of chronic cough.

DETAILED DESCRIPTION:
There is currently no national cohort study on chronic cough in China. Preliminary researches indicated heterogeneity in the clinical phenotypes and hypersensitivity associated with chronic cough, highlighting the need to establish a large chronic cough cohort for further study. The completion of this project will provide real-world data for the management of chronic cough patients, contributing to the improvement of prevention, treatment, and management standards. It will also provide Chinese data for further refining cough guidelines. Additionally, by elucidating the phenotypes and molecular subtypes related to chronic cough, this study will be significant for identifying relevant targets to guide new drug development for chronic cough. This multicenter, prospective, observational study will enroll patients with chronic cough in a real-world clinic. Baseline information including demographics, cough characteristics, past treatment history, laboratory test results, initial diagnosis and treatment details will be recorded by using an online registration and follow-up platform. After the baseline data registration, we will conduct annual follow-ups for these patients over a period of two years. The cough prognosis and medication using history will be recorded at every follow-up. Some patients will provide biological samples such as sputum supernatant, serum, etc at baseline and follow-up. The diagnosis and treatment process for these patients is based on clinical practice/guideline standards, without any other interventions.

ELIGIBILITY:
Inclusion Criteria:

* Is over 18 years old
* Cough as the sole or main symptom
* Has cough lasting more than 8 weeks
* No obvious findings of Chest X-ray / Chest CT
* Has no other evident diagnoses (e.g. IPF, NCFB, COPD, bronchiectasis, lung cancer)
* Has given signed consent for inclusion in the study

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic cough visiting the respiratory clinic or hospitalized.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline demographics, clinical and pathophysiologic characteristics of the total patients in the chronic cough cohort | After 6000 patients entry at baselin
  The demographics, and clinical characteristics included age, sex, BMI, smoking history, cough triggers, cough timing, cough complications and associated symptoms, comorbidities, previous treatment and response, cough severity outcomes evaluated by questionnaires including cough VAS, urge to cough VAS, CET, LCQ. Blood eosinophils counting, lung function and FeNO measurements were performed and recorded.
The prognosis of chronic cough in a real-word clinic | From baseline to the end of follow-up at the second year
  Elucidating the prognosis of the total patients after 2 yeas follow-up. Cough relief will be reported by patients-self and risk factors for patients with persistent cough will be investigated. After 2 years from the baseline, patients will be visited at clinic or through telephone, cough VAS, urge to cough VAS, CET and LCQ will be completed. Identifying the risk factors for patients with persistent cough by analyzing the demographic information and baseline clinical characteristics including cough duration, comorbidities, accompanying symptoms, airway inflammation biomarkers and treatment situations during the follow-up period, etc.
Identifing phenotypes and endotypes, based on biomarkers and/or clinical parameters. | After baseline entry and At the first or second year follow-up
  To elucidate the potential phenotypes and endotypes of chronic cough, demographics, baseline clinical characteristics including cough duration, cough triggers, cough timing, cough complications and associated symptoms, comorbidities etc., cough severity evaluated by cough VAS, urge to cough VAS, CET and LCQ and baseline diagnostic tests including lung function, FeNO, blood routine tests will be analyzed. Cough relief status also will be recorded during the annual follow-up. Further more, biological samples including peripheral blood mononuclear cells (PBMC), serum, sputum samples including sputum supernatant, sputum cells and urine were collected from a subset of patients at baseline and at the 1-year follow-up. For some patients with refractory chronic cough, additional biological specimens such as airway mucosa and bronchoalveolar lavage fluid will be collected. These samples will undergo transcriptomics, metagenomics, proteomics, metabolomics, whole exome sequencing, single-cell AT

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Lai, PhD, Principal Investigator — The First Affliated hospital of Guangzhou Medical University
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China